CLINICAL TRIAL: NCT02234427
Title: Pharmacogenomics of Antiplatelet Response
Acronym: PARes-III
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rehan Qayyum, Assistant Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PARes-III
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis
Keywords: aspirin, atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aspirin (Experimental)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 2-week aspirin therapy (81mg/day)

SUMMARY:
This clinical trial will examine with effect of 2-week aspirin therapy on platelet gene expression in persons at high-risk of developing heart attacks due to family history of early-onset coronary artery disease

DETAILED DESCRIPTION:
In this clinical trials we will select individuals from GeneSTAR cohort based o their platelet function. Equal number of individuals will be selected from each race and gender and from low or high platelet aggregation. We will have baseline platelet functions performed and baseline platelet gene expression examined. Participants will be given 2-week supply of aspirin(81 mg/daily) and will be examined at the end of 2-weeks with platelet aggregation studies and a repeat platelet gene-expression (using RNA-seq). The ultimate goal is to examine platelet gene expression differences due to aspirin and across different gender, race, platelet-aggregation groups.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 years
* GeneSTAR participant
* No personal History of Coronary Artery Disease
* Women who are post-menopausal
* Women who are using a reliable method of contraception, such as history of tubal ligation, IUD or taking OCP

Exclusion Criteria:

* Taking aspirin prescribed by physician
* weight < 60 kg
* History of recent or current bleeding
* allergy to aspirin or history of adverse events to aspirin
* serious comorbid conditions (such as AIDS, active cancer)
* high blood pressure (>160/95)
* History of gastrointestinal ulcer/bleeding
* Mental incompetence to make decision to participate.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rehan Qayyum, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- See also: GeneSTAR Research Program — http://www.genestarstudy.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin
Started | 34
Completed | 33 (One individual withdrew after first visit)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.3)
Gender [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  African Americans | 17
  Caucasians | 17

OUTCOME MEASURES:

1. Primary Outcome: Differential Gene Expression
Description: Differences in platelet transcriptome before and after 2-week aspirin therapy The expression levels of genes before aspirin therapy was compared with the expression level of the genes after aspirin therapy. The expression levels were measured using the FPKM unit (Fragments Per Kilobase of transcript per Million mapped reads). The gene with the highest difference (pre vs. post) in FPKM is being reported with name in the units area and the actual difference in the number area
Time Frame: 2-weeks
Population: The data were analyzed combining results from two studies (24 from this study and additional 33 individuals from study NCT01894555; total population size = 57) to improve the power to detect a difference. Same results are reported for the two studies. Note that the top most gene (HBG1) with the lowest p-value is being reported.
Measure: Mean (Standard Error); unit: FPKM for HBG1 Gene
Arm/Group | Aspirin
Number analyzed (Participants) | 57
FPKM for HBG1 Gene | 77.1 (19.8)
Statistical Analysis 1: Comparison: Aspirin; Null Hypothesis: There is no difference in gene expression before and after aspirin therapy; Test type: Superiority or Other; p < 0.000005, negative binomial — Above noted p-value is adjusted for multiple comparisons. Analysis was performed using the TopHat/Cufflinks pipeline. The differential expression algorithm uses a beta distribution and the overdispersion with a negative binomial distribution

ADVERSE EVENTS:
Arm/Group | Aspirin
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No